

A Phase 1b, open-label, boost-optimization study of an adenoviral-**Protocol Title:** 

vector based oral norovirus vaccine (VXA-G1.1-NN) expressing GI.1

VP1 administered orally to healthy adult volunteers

**Protocol Number:** VXA-NVV-105

**Protocol Version, Date:** Original v1.0, 31-MAR-2021

**ICON GPHS ID:** 4559-0016

**Document Version, Date:** Final v2.0, 18-AUG-2021

Prepared by: Chang Liu, PhD

Senior Biostatistician

On behalf of: Vaxart Biosciences, Inc.

170 Harbor Way, Suite 300

South San Francisco, CA 94080

#### Confidentiality statement:

- The information provided in this document is strictly confidential.
- The recipients of the SAP must not disclose the confidential information contained within this document or any related information to other persons without the permission of the sponsor.
- In addition, the recipient of the SAP must keep this confidential document in a controlled environment which prevents unauthorized access to the document.



## Signature Page

| Prepared at ICON GPHS by: | |
|--------------------------------------------------|--------|
| Chang Liu, PhD | |
| Senior Biostatistician | |
| <br>Signature | Date |
| o.g | 2 4.10 |
| Approved at ICON GPHS by: | |
| Toana Kawashima, MS | |
| Manager, Biostatistics | |
| Signature | Date |
| Approved at Vaxart Biosciences by: | |
| Shanita Crawford | |
| Senior Global Clinical Trials Manager | |
| Signature | Date |
| Consulting Biostatistician at Vaxart Biosciences | |
| Jeffery A. Davidson, PhD | |
| Signature | Date |



## **Revision History**

| Version | Date | Revisions |
|---|---|---|
| 0.1 | 15-APR-2021 | Initial draft |
| 0.2 | 21-APR-2021 | Revised draft after incorporating internal comments. |
| 0.3 | 30-APR-2021 | Revised draft after incorporating sponsor's comments. |
| 1.0 | 03-MAY-2021 | Finalized SAP after sponsor review. |
| 1.1 | 23-JUL-2021 | Revised SAP to incorporate analysis (responder analysis and ANCOVA) for immunogenicity endpoints and some additional internal comments. |
| 2.0 | 18-AUG-2021 | Finalized SAP after reviewing and accepting sponsor's edits and comments. |



## **Contents**

| 1.0 | Introduction | 8 |
|---|---|---|
| 2.0 | Study Objectives | 8 |
| 2.1 | Primary objective | 8 |
| 2.2 | Secondary objective | |
| 2.3 | Exploratory objectives | 8 |
| 2.4 | Safety objectives | 8 |
| 3.0 | Study Design | 8 |
| 3.1 | General study design | 8 |
| 3.2 | Randomization and blinding | 9 |
| 3.3 | Study treatments and assessments | 9 |
| 4.0 | Study Endpoints | 13 |
| 4.1 | Primary endpoints | 13 |
| 4.2 | Secondary endpoints | 13 |
| 4.3 | Exploratory endpoints | 13 |
| 5.0 | Sample Size and Power | 14 |
| 6.0 | Analysis Populations | 14 |
| 6.1 | Full Analysis Set (FAS) | 14 |
| 6.2 | Safety population (Safety) | 14 |
| 6.3 | Per-Protocol population (PP) | 14 |
| 6.4 | Protocol deviations/violations and exclusions from analysis sets | 14 |
| 7.0 | Statistical Considerations and Analysis | 15 |
| 7.1 | Derived Variables | 15 |
| 7.2 | Handling of missing data and outliers | 16 |
| 7.3 | Missing data analysis methods | 16 |
| 8.0 | Statistical Methods | 17 |
| 8.1 | General statistical conventions | 17 |
| 8.2 | Subject disposition | 17 |
| 8.3 | Protocol deviations | 18 |
| 8.4 | Demographics and baseline characteristics | 18 |
| 8.4.1 | Demographics | 18 |
| 8.4.2 | Baseline and disease characteristics | 18 |
| 8.4.3 | Medical history | 18 |
| 8.4.4 | Prior and concomitant medications | 18 |



| 8.5 | Extent of exposure | 19 |
|-------|-----------------------------------------------------------------|----|
| 8.6 | Immunogenicity analysis | 19 |
| 8.6.1 | 1 Analysis methods | 19 |
| 8.6.1 | 1.1 Responder Analysis | 20 |
| 8.6.1 | 1.2 Analysis of Covariance (ANCOVA) | 20 |
| 8.6.2 | 2 Multiplicity | 20 |
| 8.6.3 | Treatment by center interaction analysis (multi-center study) | 20 |
| 8.7 | Safety analysis | 20 |
| 8.7.1 | 1 Adverse events | 21 |
| 8.7.2 | 2 Clinical laboratory evaluations | 22 |
| 8.7.3 | 3 Vital signs | 22 |
| 8.7.4 | Physical examinations | 22 |
| 8.7.5 | 5 Other safety assessments | 23 |
| 8.8 | Follow-up Period Analysis | 23 |
| 9.0 | Changes to Planned Analysis from Study Protocol | 23 |
| 10.0 | References | 23 |
| 11.0 | Appendices | 23 |
| Appe | endix 1 - Grading of Solicited Symptoms of Reactogenicity | 24 |
| Appe | endix 2 – Grading of Laboratory Abnormalities (Serum Chemistry) | 25 |
| Appe | endix 3 – Grading of Laboratory Abnormalities (Hematology) | 26 |
| Appe | endix 4 – Grading of Laboratory Abnormalities (Urinalysis) | 27 |

Version: Final v2.0, Date: 18-AUG-2021



## **List of Abbreviations**

| Abbroviction | Funlanation |
|--------------|----------------------------------------------|
| Abbreviation | Explanation |
| Ad5 | Adenovirus type 5 |
| AECL | Adverse event |
| AESI | Adverse event of special interest |
| ALT | Alanine transaminase |
| ANCOVA | Analysis of covariance |
| ATC | Anatomical therapeutic chemical |
| ASC | Antibody secreting cells |
| AST | Aspartate aminotransferase |
| BMI | Body mass index |
| BT50 | Blocking titer 50 |
| BUN | Blood urea nitrogen |
| СРК | Creatine phosphokinase |
| CRF | Case report form |
| CSR | Clinical study report |
| DIC | Disseminated intravascular coagulation |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| ELISA | Enzyme-linked immunosorbent assay |
| ELISpot | Enzyme-linked immune absorbent spot |
| EOS | End of study |
| ER | Emergency room |
| ET | Early termination |
| FAS | Full analysis set |
| GCP | Good clinical practices |
| GM | Geometric mean |
| GMFR | Geometric mean fold rise |
| GMT | Geometric mean titer |
| GPHS | Government & Public Health Solutions |
| HBGA | Histo-blood group antigen |
| HBsAg | Hepatitis B surface antigen |
| HCV | Hepatitis C virus |
| HIV | Human immunodeficiency virus |
| ICH | International Council for Harmonization |
| IgA | Immunoglobulin A |
| IgG | Immunoglobulin G |
| IQR | Interquartile range |
| IU | International units |
| LS-GMR | Least square geometric mean ratio |
| LSM | Least square mean |
| MedDRA | Medical dictionary for regulatory activities |
| MSD | Meso scale discovery |
| NOCI | New onset of chronic illness |
| PBMC | Peripheral blood mononuclear cells |
| PI | Principal investigator |
| PP | Per protocol |
| PT | Prothrombin time |
| PTT | Partial thromboplastin time |
| SAE | Serious adverse event |
| U/L | Conodo davordo event |



| Abbreviation | Explanation |
|--------------|------------------------------|
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SI | Standard international |
| SOC | System organ class |
| SoE | Schedule of Events |
| TLF | Tables, listings and figures |
| ULN | Upper limit of normal |
| VP1 | Vaccine protein 1 |
| WBC | White blood cell |



#### 1.0 Introduction

The purpose of this Statistical Analysis Plan (SAP) is to provide detailed descriptions of the statistical methods, data derivations, and data displays for the study protocol VXA-NVV-105 Original "A Phase 1b, open-label, boost-optimization study of an adenoviral-vector based oral norovirus vaccine (VXA-G1.1-NN) expressing GI.1 VP1 administered orally to healthy adult volunteers" dated 31-MAR-2021 for final analysis. The table of contents and templates for the table, listing and figures (TLFs) will be produced in a separate document.

Any deviations from this SAP will be described and justified in the Clinical Study Report (CSR).

The preparation of this SAP has been based on International Council for Harmonisation (ICH) E9 and Good Clinical Practice (GCP) guidelines.

All data analyses and generation of TLFs will be performed using SAS 9.4® (or higher).

## 2.0 Study Objectives

#### 2.1 Primary objective

To evaluate the immunogenicity of VXA-G1.1-NN with repeat-dose administration at Day 1 and varying boost schedules (Week 4, 8 or 12 post initial dose) in healthy adults aged 18-55, inclusive.

#### 2.2 Secondary objective

To assess the safety and tolerability of VXA-G1.1-NN with repeat-dose administration at varying boost schedules (Week 4, 8 or 12) in healthy adults aged 18-55, inclusive.

#### 2.3 Exploratory objectives

- To assess additional safety parameters
- To assess long-term safety of VXA-G1.1-NN through 6 months after last vaccination
- To assess additional immunogenicity parameters of VXA-G1.1-NN

#### 2.4 Safety objectives

Safety objectives are included as part of the secondary and exploratory objectives.

#### 3.0 Study Design

#### 3.1 General study design

This is a Phase 1b, open-label, boost-optimization study to evaluate the immunogenicity, safety and tolerability of VXA-G1.1-NN with repeat-dose administration at Day 1 and varying boost schedules in healthy



adult subjects aged 18-55. Thirty subjects will be enrolled to one of the three treatment cohorts (10 subjects in each cohort) with varying boosting vaccination schedules at Week 4, 8 or 12, respectively, post the initial vaccination on Day 1 such that each subject will receive two doses of  $1\times10^{10}$  IU  $\pm$  0.5 log in total. See study protocol Section 5 for inclusion and exclusion criteria.

On Day 1, participants will be enrolled sequentially in order of eligibility. Participants may be assigned to cohorts based on their availability for the second dose (boost). Cohorts 3 and 2 will be enrolled prior to Cohort 1 to optimize the overall study timeline.

Table 1: Treatment Arm, Doses and Sample Sizes

| Group | Study Drug | Dose<br>(IU ±0.5 log) | Doses | Dosing Schedule | Subjects |
|---|---|---|---|---|---|
| Cohort 1 | VXA-G1.1-NN | 1x10 <sup>10</sup> | 2 | Day 1 & Week 4 | 10 |
| Cohort 2 | VXA-G1.1-NN | 1x10 <sup>10</sup> | 2 | Day 1 & Week 8 | 10 |
| Cohort 3 | VXA-G1.1-NN | 1x10 <sup>10</sup> | 2 | Day 1 & Week 12 | 10 |
| | | | | Total | 30 |

The study will include a Screening period, Study Period 1, Study Period 2, and a Follow-up Period:

- Screening Period (Day -45 to -1)
- Study Period 1 (Day 1 to 4 weeks post initial vaccination)
- Study Period 2 (4 weeks from the second vaccination: Week 4 to Week 8 for Cohort 1; Week 8 to Week 12 for Cohort 2; Week 12 to Week 16 for Cohort 3)
- Follow-up Period (6 months post the second vaccination for each cohort: Month 7 for Cohort 1,
   Month 8 for Cohort 2 and Month 9 for Cohort 3)

#### 3.2 Randomization and blinding

As VXA-NVV-105 is a Phase 1b, open-label, boost-optimization study to determine the immunogenicity, safety and tolerability of vaccine VXA-G1.1-NN at dose level  $1 \times 10^{10}$  IU  $\pm$  0.5 log with varying boosting schedules, neither randomization nor blinding will be applicable for this study. Both subjects and investigators will be aware of individual treatment assignment.

#### 3.3 Study treatments and assessments

Subject participation will last for about 7 months for Cohort 1 (4-week boost vaccination), 8 and 9 months for Cohorts 2 and 3 respectively (Cohort 2: 8-week boost vaccination; Cohort 3: 12-week boost vaccination). Subjects will be followed for 4 weeks after each dose, and through 6 months following the boosting dose. Following confirmation of eligibility during the screening period, subjects will be enrolled and receive their first



dose of study vaccine on Day 1 and their second dose of study vaccine on Day 29, Day 57 or Day 85 depending on their assigned cohort if deemed eligible after pre-dose safety assessments.

Subjects will record any potential symptoms of reactogenicity daily for 1 week after each dose and return to the site to have safety assessments and samples collected for evaluation of immunogenicity. Subjects deemed ineligible for the second vaccination due to acute illness or new medical condition may be reassessed and have a delayed second vaccination within 1 week of their scheduled vaccination visit if the condition resolves. If a subject remains ineligible after the re-assessment, they will complete an Early Termination (ET) visit and then enter the scheduled follow-up period per cohort assignment as outlined in the schedule of events (SoE). All subjects will enter the follow-up period 4 weeks after their last vaccination and will be monitored for serious adverse events (SAEs), adverse events of special interest (AESIs) and new onset of chronic illness (NOCI) through the End of Study. Subjects will also have samples collected for evaluation of immunogenicity as scheduled in SoE.

A detailed description of procedures and assessments to be conducted during the active period of this study is summarized in the Schedule of Events in Table 2 below, with those during the follow-up period summarized in Table 3.



Table 2 – Schedule of Events (Active Period)

| | - C | G. I. D. | 11 61 41 | | e Period | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Screen | Study Period | l 1 – Cohorts 1 | | | | | | | |
| | | | | Stud | y Period 2 – ( | | | | | |
| | | | | | | Study Peri | iod 2 – Cohor | | | |
| | | | | | | | | · | iod 2 – Cohort 3 | |
| Study Day | -45d to<br>-1 d | Day 1<br>(Wk 0) | Day 8<br>(Wk 1) | Day 29<br>(Wk 4) | Day 36<br>(Wk 5) | Day 57<br>(Wk 8) /ET <sup>1</sup> | Day 64<br>(Wk 9) | Day 85 (Wk<br>12)/ET <sup>2</sup> | Day 92<br>(Wk 13) | Day 113<br>(Wk16)/ET <sup>3</sup> |
| Visit Window (days) | | n/a | 0 | ±2 | 0 | ±2 | 0 | ±2 | 0 | ±2 |
| Informed consent | X | | | | | | | | | |
| Inclusion/Exclusion | X | X | | X | | | | | | |
| Demographics | X | | | | | | | | | |
| Medical history | X | | | | | | | | | |
| Stool for occult blood | X | | | | | | | | | |
| Blood Sample (HBsAg, HCV, HIV) | X | | | | | | | | | |
| Urine drug screen | X | | | | | | | | | |
| Serum Pregnancy Test <sup>a</sup> | X | X | | x1 | | x <sup>2</sup> | | X <sup>3</sup> | | |
| Physical examination | X | Xb | Xb | Xb | Xb | Xb | хb | Xb | Xb | Xp |
| Vital Signs | X | X | X | X | X | X | X | X | X | X |
| Safety laboratory tests | X | X <sup>c</sup> | X | X | X | X | X | X | X | X |
| Urinalysis | X | X | X | X | X | X | X | X | X | X |
| COVID vaccination status | X | | | | | | | | | |
| Vaccination | | X | | X1, d,e | | X,2, d,e | | x <sup>3</sup> , d,e | | |
| Dispense Solicited Symptom Diary | | x1,2,3 | | x1 | | $x^2$ | | X <sup>3</sup> | | |
| Review & Collect Solicited Symptom Diary | | | X | | x <sup>1</sup> | | x <sup>2</sup> | | X <sup>3</sup> | |
| Review prior & concomitant medication | X | X | X | X | X | X | X | X | X | X |
| Query for AEs, SAEs, AESIs andNOCIs | | X | X | X | $X^{1,f}$ | X <sup>1,f</sup> | $X^{2,f}$ | X <sup>2,f</sup> | X <sup>3,f</sup> | X <sup>3,f</sup> |
| ample Collection Immunogenicity Assessment | s | | | | | | _ | | - | • |
| Serum | | X1,2,3g | | x1,2,3 | | x <sup>1,2</sup> | | x <sup>2,3</sup> | | x <sup>3</sup> |
| Whole blood (Flow-Based) | | x1,2,3 | x1,2,3 | x <sup>1</sup> | x <sup>1</sup> | $X^2$ | x <sup>2</sup> | X <sup>3</sup> | X <sup>3</sup> | |
| Whole blood (PBMC) | | x1,2,3 | x1,2,3 | x <sup>1</sup> | x <sup>1</sup> | x <sup>2</sup> | x <sup>2</sup> | X <sup>3</sup> | x <sup>3</sup> | |
| Nasal Swab (Sam Device) | | x1,2,3 | | x1,2,3 | | x <sup>1,2</sup> | | x <sup>2,3</sup> | | x <sup>3</sup> |
| Saliva Sample | | X1,2,3 | | x1,2,3 | | x <sup>1,2</sup> | | X <sup>2,3</sup> | | X <sup>3</sup> |



#### Table 3 – Schedule of Events (Follow-up Period)

| | | F | ollow-Up Period | | | |
|---|---|---|---|---|---|---|
| | ( | COHORT 1 | COI | HORT 2 | COHORT 3 | |
| Study Day | Months 3, 4, 5, 6 | Month 7 (Wk 28)/ EOS | Months 4, 5, 6, 7 | Month 8 (Wk 32)/EOS | Months 5, 6, 7, 8 | Month 9 (Wk 36)/EOS |
| Telephone Visit | X | | X | | X | |
| Visit Window (days) | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 |
| Query for SAEs, AESIs and NOCIs | X | X | X | X | X | X |
| Sample Collection Immunogenicity Asses | sments | | | | | |
| Serum | | X | | X | | X |
| Whole blood (PBMC) <sup>a</sup> | | X | | X | | X |
| Nasal Swab (Sam Device) | | X | | X | | X |
| Saliva | | X | | X | | X |

AE, adverse event; AESI, Adverse event of special interest; EOS, End of Study; ET, Early Termination; HCV, Hepatitis C Virus; HIV, Human Immunodeficiency Virus; NP, Nasopharyngeal; NOCI, New Onset of Chronic Illness; PBMC, peripheral blood mononuclear cells; SAE, serious adverse event.

BST1302-SOP-T01/v1.0/2020 Page 12 of 27

 $<sup>^{1}</sup>$  = Cohort 1;  $^{2}$  = Cohort 2;  $^{3}$  = Cohort 3.

<sup>&</sup>lt;sup>a</sup> For women of childbearing potential. Test at Day 1 and at second dose (boost). Test at 2<sup>nd</sup> Study drug administration visit can be serum or urine test.

b Targeted.

<sup>&</sup>lt;sup>c</sup> If screening lab tests are performed within 2 days prior to dosing, no need to repeat at Day 1.

d Assess eligibility to receive second dose. Participants with acute illness or new medical condition may be re-assessed, and if the condition resolves, have a delayed 2<sup>nd</sup> dose within 1 week of scheduled visit.

e If participants are not eligible to receive their 2<sup>nd</sup> dose, they immediately enter the follow-up period.

f AEs will only be collected for 4 weeks following each study drug administration.

g An aliquot of serum collected at baseline will be stored for testing (e.g. Platelet Factor 4 [PF4] antibody ELISA) should an AESI related to blood clots be reported anytime during the study period.

a Optional.



### 4.0 Study Endpoints

#### 4.1 Primary endpoints

- Number of VP1 specific IgA antibody secreting cells (ASC) by enzyme-linked immunospot (ELISpot) by treatment group and visit
- Geometric mean titer (GMT) and geometric mean fold rise (GMFR) over the initial GMT of Norovirus
   G1.1 histo-blood group antigen (HBGA) blocking antibodies (BT50) by treatment group and visit
- Geometric mean (GM) and GMFR over the initial results of VP1 specific serum IgG by Meso Scale
   Discovery (MSD) by treatment group and visit

#### 4.2 Secondary endpoints

- Frequencies, durations, and severities of solicited symptoms of reactogenicity (local, systemic) for 1
  week following each dose of study drug by treatment group
- Frequencies, durations, and severities of unsolicited AEs, SAEs, AESIs and NOCIs through each
  active study period (4 weeks post each vaccination) by treatment group
- Number and percentages of subjects with ≥2-, 3-, 4-fold increase over baseline titer of Norovirus
   G1.1 HBGA BT50 results by treatment group and visit
- Geometric Least Square Mean (LSM) of post-dose Norovirus G1.1 HBGA BT50 titer by treatment group and visit adjusted for baseline titer level
- Least Square Geometric Mean Ratio (LS-GMR) of post-dose titer Norovirus G1.1 HBGA BT50 between treatment groups by visit adjusted for baseline titer level

#### 4.3 Exploratory endpoints

- Frequencies of clinically significant abnormalities in laboratory parameters (chemistry, hematology and urinalysis) at 1 week after each study drug dose and in vital signs immediately following each dose by treatment group
- Frequencies, durations, and severities of all SAEs, AESIs and NOCIs through 6 months after the last vaccination by treatment group
- The following additional immunogenicity parameters will be analyzed by treatment group and visit, and will be reported in the CSR:
  - o Number of VP1 specific IgG ASC
  - GM and GMFR over the initial results of VP1 specific serum IgA

Additional exploratory immunogenicity assays not listed above may also be performed to further evaluate the activity of the VXA-G1.1-NN vaccine candidate. The data from such exploratory assays will be reported outside the scope of this SAP.



### 5.0 Sample Size and Power

No formal sample size calculation was performed for the study. Thirty subjects in total (10 in each cohort) are planned to be enrolled based on experience of a typical Phase I vaccine study.

#### 6.0 Analysis Populations

#### 6.1 Full Analysis Set (FAS)

The FAS will consist of all subjects who have received at least one dose of vaccine VXA-G1.1-NN. Subjects will be included in the analysis according to the cohort to which they are assigned. Subjects who have been enrolled but never received the study vaccine will be excluded from the analysis.

#### 6.2 Safety population (Safety)

Safety population will consist of all subjects who receive at least one dose of study vaccine and will be analyzed according to the cohort to which they belong according to the actual dosing schedule. Subjects who have been enrolled but never received the study vaccine will be excluded from the analysis.

#### 6.3 Per-Protocol population (PP)

The per-protocol population will consist of all subjects in the FAS who received both vaccine doses and are free from major protocol violations that warrant exclusion. Subjects will be included in the analysis according to the cohort to which they are assigned.

#### 6.4 Protocol deviations/violations and exclusions from analysis sets

All violations and exclusions of subjects from analysis sets will be identified and documented prior to data base lock and final analysis, through clinical review input provided by the sponsor, using the following sources of information:

- Supportive subject listings provided by the ICON GPHS statistician based upon data recorded in the
  CRE
- Protocol deviation logs provided by the site
- Protocol deviation listings provided by the Sponsor

Deviations from the protocol will be classified as to whether or not they are Major Deviations.

The major protocol deviations to be identified and to be included in the body of the CSR will include the following at a minimum, as well as others classified as key during review of all deviations observed:

- Failure to obtain informed consent
- Incorrect dose of vaccine
- Failure to meet eligibility criteria at baseline



## 7.0 Statistical Considerations and Analysis

#### 7.1 Derived Variables

The below table provides the list of derived variables for demographic and baseline characteristics, various duration derivations, baseline derivation and other important derivations applicable for this study.

**Table 4: Derived Variables** 

| Variables | Formula |
|---|---|
| Demographic and Baseline Charac | Demographic and Baseline Characteristics |
| Age at informed consent (in years) | Integer ((date of informed consent – date of birth + 1) / 365.25) |
| Body Mass Index | Weight (kg) / height (m) <sup>2</sup> |
| Derivation of Durations | |
| Study day at any visit | Date of interest – date of first dose of vaccine. One day is added if the difference is ≥ 0. |
| Duration of any events | End date of event – start date of event + 1 |
| Baseline Derivations | |
| Laboratory baseline | The baseline value is defined as the last observation prior to or on the date of the first dose of study drug. |
| Change from baseline | Post baseline value – baseline |
| Percent change from baseline | [(Post baseline value – baseline) / baseline] * 100 |
| Change from previous visit | Current value – previous value |
| Percent change from previous visit | [(Current value – previous value) / previous value] * 100 |
| Other Derivations | |
| Geometric mean/geometric, mean titer/geometric mean concentration | Individual values will be transformed via the natural log, mean values along with 95% CIs will be calculated, which will be transformed back to the original scale via exponentiation. |
| Geometric mean fold rise | The mean values and 95% CIs of the log ratio of post dose assay values relative to baseline will be calculated, then transformed back to the original scale via exponentiation. |
| Geometric least square mean | Least square means and 95% CIs for each treatment group will be calculated from ANCOVA with immunogenicity assay result on log scale at post dose visit as a dependent variable, treatment group as a factor and baseline immunogenicity assay result on log scale as a covariate, which will be then transformed to the original scale via exponentiation. |
| Least square geometric mean ratio | Least square mean differences and 95% CIs among treatment groups will be estimated from the abovementioned ANCOVA model, which will be then transformed to the original scale via exponentiation. |



#### 7.2 Handling of missing data and outliers

The extent and pattern of missing data for primary, secondary, and exploratory endpoints will be summarized by cohort and visit date with frequencies and percentages. No imputations will be conducted for missing data other than dates. No outliers will be eliminated.

#### 7.3 Missing data analysis methods

#### Imputation rules for missing or partial adverse event start/stop dates

- If the AE start date day is missing (month and year provided) then set the date to the first of the month, unless the month and year are the same as the first dose of study drug. In this case, set the date to the date of first dose.
- If the AE start date month is missing (year is provided) then set the month and day to January 1, unless the year is the same as the year of the first dose. In this case, set the date to the date of first dose.
- If the AE end date day is missing (month and year provided) then set the date to the last day of the month.
- If the AE end date month is missing (year is provided) then set the date to December 31 or current date, whichever is earlier.
- If the year of the AE start date or AE end date are missing, then a query to the site must be made to gather additional information. If the end date and start date are both missing, then no imputation will be done. If the start date remains missing but the end date is before first dose date, then the AE will be considered before treatment and it will not be recorded as an AE in CRF but included as medical history. If the end date is after the first dose, then the AE will be considered to have been treatment emergent.

#### Imputation rules for missing or partial medication start/stop dates

#### Start Date:

- If only day is missing, use the first day of the month.
- If day and month are missing, use the first day of the year.
- If day, month, and year are missing use the first day of the year with the same year as the first dose.

#### End Date:

- If only day is missing, use the last day of the month.
- If day and month are missing, use the last day of the year.
- If day, month, and year are missing assign 'continuing' status to the stop date.



#### 8.0 Statistical Methods

#### 8.1 General statistical conventions

All statistical procedures will be completed using SAS version 9.4 (or higher).

Continuous variables will be summarized using descriptive statistics, including number of subjects (n), mean, median, standard deviation (SD), interquartile ranges (IQR), minimum, and maximum.

For categorical variables, summaries will include counts of subjects and percentages. Percentages will be rounded to one decimal place.

For summary purposes, baseline will be defined as the last available pre-dose value. All summaries will be presented by treatment group, unless otherwise specified.

Immunogenicity titer data will be summarized using GMT/GMC and GMFR over baseline GMT/GMC. Immunogenicity data below the lower limit of quantification (LLOQ) will be summarized as LLOQ/2 in all relevant tables and will be displayed in listings in the format of source data. Immunogenicity data above the upper limit of quantification (ULOQ) will be summarized using ULOQ in all relevant tables and will be displayed in listings in the format of source data.

All subject data, including those derived, will be presented in individual subject data listings. Unless otherwise stated, unscheduled visit results will be included in date/time chronological order, within patient listings only. All listings will be sorted by subject ID, treatment group, study visit. Subject's sex and age will be also stated on each listing. Unless otherwise stated, data listings will be based on FAS.

Unscheduled data points will not be used in any summary tables separated by visit.

#### 8.2 Subject disposition

Subject disposition information will be summarized by treatment group and overall. The number and percentage of subjects who are enrolled, who are eligible/ineligible to receive the second dose of vaccine, who complete the active period of the study, and who withdraw early from the study will be presented.

The primary reasons for ineligibility and early withdrawal will also be tabulated.

The number of subjects enrolled will be used as the denominator for the percentage calculation. Subject disposition will be listed.

The number and percentage of subjects in each analysis set will also be tabulated. A listing of each subject excluded from an analysis population will be listed as well as the reason why they were excluded from the population.



#### 8.3 Protocol deviations

The number of subjects excluded from FAS, Safety, and Per-protocol analysis sets and reasons for exclusion will be summarized by treatment group and overall.

Population membership details will be listed, including reason for exclusion from each population.

Protocol deviation data are not captured in the clinical database and therefore will not be reported on individually within the scope of the SAP. Protocol deviations will be summarized in the final CSR.

#### 8.4 Demographics and baseline characteristics

#### 8.4.1 Demographics

Summary of demographics will be based on the FAS. Age at consent in years, height in cm, weight in kg and BMI (kg/m²) will be summarized descriptively using mean, SD, median, IQR, and range. Sex at birth, race and ethnicity will be summarized using frequencies and percentages.

#### 8.4.2 Baseline and disease characteristics

The baseline continuous characteristics (vital signs) will be summarized descriptively for the safety population using mean, SD, median, IQR, and range. The baseline categorical characteristics (results of physical exam, chemistry, hematology and urinalysis) will be summarized (normal vs abnormal) using frequencies and percentages for the safety population.

#### 8.4.3 Medical history

A summary of medical history will be presented by system organ class (SOC) and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA) version 24.0 by cohort at baseline.

#### 8.4.4 Prior and concomitant medications

Medications used in this study will be coded by using the World Health Organization Drug Dictionary Enhanced (WHODrug version March 1, 2021).

Concomitant medication is defined as any prescription or over-the-counter preparation. Use of concomitant medication from 4 weeks before Day 1 through 4 weeks after the last dose administration must be recorded in eCRF from the subject's medical file along with reason for use, dates of administration including start and end dates, dosage information including dose and frequency. Medications for pre-existing medical conditions or required for a medical condition during the study are allowed if not considered exclusionary. Medications specifically prohibited in the exclusion criteria (Section 5.2 in study protocol) are not allowed during the active study period, unless deemed medically necessary by the investigator. The Sponsor's medical monitor (or designee) should be contacted if there are any questions regarding concomitant or prior medications.



Concomitant medications will be summarized descriptively using frequency tables by Anatomical Therapeutic Chemical (ATC) class (hierarchically by Level I, II and III) and cohort in the descending order of overall frequency. All concomitant medications will be presented in listings as well.

Details for imputing missing or partial start and/or stop dates of medication are described in Section 7.3.

### 8.5 Extent of exposure

Vaccines will be administered on-site for all subjects. All subjects will receive the first dose on Day 1. Subjects will receive the second dose on Day 29 for Cohort 1 (4-week boost vaccination), Day 57 for Cohort 2 (8-week boost vaccination), and Day 85 for Cohort 3 (12-week boost vaccination), respectively, allowing for a potential delay up to 1 week. Frequencies and percentages will be calculated for the number of doses received (1 dose or 2 doses), the presence of delay in administering the second dose, whether vaccination is administered per protocol along with reasons why vaccine administration is not per protocol.

#### 8.6 Immunogenicity analysis

This section addresses the analysis methods for immunogenicity outcomes.

#### 8.6.1 Analysis methods

Immunogenicity will be evaluated using cellular and humoral immune function assays from blood and mucosal (saliva and nasal swab) samples. Samples will be collected from all subjects according to the time points specified in the SoE.

Results of the following immunogenicity assay results will be summarized descriptively by treatment group and visit and will be reported in the final CSR. Specific endpoints are listed in Sections 4.1 and 4.3.

- VP1 specific IgA ASC by ELISpot
- Norovirus G1.1 HBGA BT50
- VP1 specific serum IgG by ELISA or MSD
- VP1 specific IgG ASC by ELISpot
- VP1 specific serum IgA by ELISA or MSD

Additional exploratory endpoints will be evaluated and reported outside the scope of this SAP.

Kolmogorov-Smirnov test will be used to examine the normality assumptions of the immunogenicity assay results in log scale for each treatment group. If normality assumptions are met for all treatment groups, pairwise comparisons will be performed between treatment groups using Student t-test; Wilcoxon rank sum test will be used if otherwise.



#### 8.6.1.1 Responder Analysis

A responder analysis at each appropriate post-dose follow-up visit (see Table 1 and Table 2 for specific timings) will be conducted for the Norovirus G1.1 HBGA BT50. During active period, the numbers and percentages (with 95% CIs) of subjects with a  $\geq 2$ -, 3- or 4-fold increase from baseline antibody levels will be summarized, respectively. Durability of immune responses will be evaluated using the safety follow-up period samples collected at 6 months post the second dose (Month 7 for Cohort 1, Month 8 for Cohort 2, and Month 9 for Cohort 3). Numbers and percentages of subjects with a  $\geq 2$ -, 3- or 4-fold increase from baseline antibody levels at both 28 day post the second dose (Day 57 for Cohort 1, Day 85 for Cohort 2, and Day 113 for Cohort 3) and 6 month post the second dose will be summarized, where percentages will be calculated as of the number of subjects with a  $\geq 2$ -, 3- or 4-fold increase from baseline antibody levels at 28 day post the second dose. Fisher's exact test will be used to compare the percentages of responders for each category among cohorts.

#### 8.6.1.2 Analysis of Covariance (ANCOVA)

To account for the potential differences in baseline antibody level, ANCOVA will be used to analyze and compare the immunogenicity endpoints at each post-dose visits conditioning on baseline values for the Norovirus G1.1 HBGA BT50 assay. Separate models will be estimated at each post-dose visit, using log titer as a dependent variable, treatment group as a factor and baseline log titer as a covariate. LSMs for each cohort and differences in LSM between cohorts will be estimated from each model along with 95% CIs. Both LSMs for each cohort and the differences in LSM between cohorts along with their 95% CIs will be exponentiated to the original scale, resulting geometric LSMs for each cohort and LS-GMR between cohorts. In order to compare immunogenicity assay results among treatment groups, significance on 28 days post the second dose will be used. If the ANCOVA demonstrates overall significance on 28 days post the second dose, pairwise comparisons will be performed.

#### 8.6.2 Multiplicity

There will be multiple outcomes pertaining to immunogenicity; however, each outcome will be analyzed separately, and no corrections will be made to account for multiplicity. Pairwise comparisons among cohorts will also be conducted; Holm-Bonferroni method will be used to control family-wise error rate, both adjusted and unadjusted p-values will be reported.

#### 8.6.3 Treatment by center interaction analysis (multi-center study)

Not applicable since this is a single-center study.

#### 8.7 Safety analysis

This section describes the safety analyses that will be conducted during the active and follow-up periods (i.e., the safety analyses on all data collected during the active and follow-up periods and all data collected in subjects who dropped-out during the active and follow-up periods).



All definitions relative to safety endpoints are detailed in Section 4.4.

Safety analyses will be conducted on the safety population and will be performed for all safety variables specified below.

All safety data will be summarized by cohort and study visit as well as by overall study population.

The safety analyses of changes from baseline to a specific time point in safety variables (e.g., vital signs) will only include subjects from the safety population who have data available at both the baseline and the time point under considerations unless otherwise specified.

#### 8.7.1 Adverse events

All adverse events (AEs) (except for solicited AEs) will be classified by primary SOC and preferred term according to the Medical Dictionary for Regulatory Activities (MedDRA) Version 24.0

AEs will be categorized by solicited AEs, unsolicited AEs (including both AESIs and NOCIs) and SAEs, where the frequencies and durations of each will be summarized by cohort, severity and relatedness to study treatment.

Solicited AEs are predefined systemic signs and symptoms of reactogenicity for which the subjects are specifically questioned; including fever (any temperature 100°F or higher), headache, myalgia (muscle pain), abdominal pain, anorexia (defined as not eating), nausea, vomiting, diarrhea and malaise/fatigue. Frequencies and percentages for each solicited symptom will be calculated. Severities of solicited AEs will be graded according Appendix 1. Definitions of AE, AESI and NOCI are provided in the study protocol (refer to Tables 7 – 11 in the study protocol Section 10.3).

Unsolicited AEs will be summarized by SOC and preferred term for AESIs and NOCIs combined where the events will be sorted by descending overall frequency within each SOC and preferred term according to the total number of events.

Frequencies and percentages of SAEs will be summarized by treatment group, along with specifics including whether the AE is associated with a congenital anomaly or birth defect, whether the AE results in persistent or significant disability or incapacity, initial or prolonged hospitalization, and death, whether the AE is lifethreatening, or medically important but not covered by other serious criteria.

The severity of AEs will be assessed by the clinician using a protocol-defined grading system. For events that are not listed in the protocol-defined grading system, refer to Table 12 in the study protocol Section 10.3 for classifying severity.

Relationships of AEs to study vaccine are categorized as not related, possibly related, probably related, and definitely related (refer to Table 17 in the study protocol Section 10.3.1 for details).

Details for imputing missing or partial start dates of adverse events are described in Section 7.2 of this SAP.



Where a subject has the same adverse event, based on preferred terminology, reported multiple times in the treatment period, the subject will only be counted once at the preferred terminology level in adverse event frequency tables.

Where a subject has multiple AEs within the same SOC in the treatment period, the subject will only be counted once at the SOC level in AE summary tables.

Listings will be provided for solicited AEs, unsolicited AEs (including both AESIs and NOCIs) and SAEs, where patient information, SOC and preferred term, durations, severities, relatedness to study treatment, outcomes, and actions will be included.

#### 8.7.2 Clinical laboratory evaluations

Clinical laboratory evaluations include serum chemistry, hematology and urinalysis. For the purposes of summarization in both the tables and listings, all laboratory values will be presented in SI units. If a lab value is reported using a nonnumeric qualifier e.g., less than (<) a certain value, or greater than (>) a certain value, the given numeric value will be used in the summary statistics, ignoring the nonnumeric qualifier. Severity of laboratory results will be categorized as mild, moderate, severe and potentially life threatening according to Appendices 2 - 4 in current document.

All laboratory data obtained between screening visit and the end of study will be used for the laboratory safety analysis. Frequencies and percentages of subjects with abnormal laboratory results will be summarized for each laboratory test and further by individual laboratory parameters at each time point. Shift tables for hematology and chemistry laboratory assessments between baseline and each subsequent visit will be provided if applicable.

Abnormal laboratory results will be listed by treatment group and visit, including patient information, lab parameter, lab results along with normal ranges, and abnormality criteria.

#### 8.7.3 Vital signs

Visit values and changes from baseline for vital sign measurements (blood pressure, oral temperature, heart rate and respiratory rate) will be summarized by cohort at each visit using descriptive statistics. Visit values will be calculated as the mean of all available measurements per parameter if multiple measurements are taken during the visit.

#### 8.7.4 Physical examinations

Physical examinations will be conducted at baseline and all subsequent visits. At baseline, a complete physical examination will be conducted and results by body system and specific abnormalities along with clinical significance will be summarized by treatment group using frequencies and percentages. At subsequent visits, targeted and symptom-directed physical examinations will be conducted. Any changes from previous physical examination will be documented; frequencies and percentages of abnormal findings



will be summarized by treatment group; if deemed as adverse events, results will be listed accordingly by subject and summarized by treatment group at each visit.

#### 8.7.5 Other safety assessments

Urine drug screen, tests for hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody types 1 and 2, stool for occult blood and alcohol screen will be administered at screening for all subjects. Women with childbearing potential will receive serum pregnancy test at screen, serum or urine pregnancy test on dosing visits. Results of the abovementioned safety assessments will be summarized via listings.

#### 8.8 Follow-up Period Analysis

Following completion of the study Active Period for all enrolled subjects, the study database will be cleaned and locked then the CSR will be finalized. Safety and immunogenicity data collected during the safety follow-up period will be appended to the CSR via an addendum after completion of the study (6 months post the last vaccination), where tables and listings pertaining to SAEs, immunogenicity endpoints will be updated accordingly incorporating data collected during the safety follow-up period.

## 9.0 Changes to Planned Analysis from Study Protocol

None.

#### 10.0 References

1. ICH E9 Statistical Principles for Clinical Trials (R1)

### 11.0 Appendices



Appendix 1 - Grading of Solicited Symptoms of Reactogenicity

| | Grading | | | | |
|---|---|---|---|---|---|
| Symptom | Normal<br>0 | Mild<br>Grade 1 | Moderate<br>Grade 2 | Severe<br>Grade 3 | Life Threatening<br>Grade 4 |
| Fever | < 100.4°F | 100.4 – 101.1°F | 101.2 – 102.0°F | 102.1 – 104°F | > 104.0°F |
| (oral temp) | (< 38.0°C) | $(38.0 - 38.4^{\circ}C)$ | $(38.5 - 38.9^{\circ}C)$ | $(39.0 - 40^{\circ}C)$ | (>40°C) |
| Headache | None | No interference<br>with activity | Repeated use of<br>nonnarcotic pain<br>reliever > 24 hours<br>or some interference<br>with activity | Significant; any use<br>of narcotic pain<br>reliever or prevents<br>daily activity | ER visit or<br>hospitalization |
| Myalgia | None | Easily tolerated,<br>causing minimal<br>discomfort and<br>does not interfere<br>with everyday<br>activities <sup>a</sup> | Sufficiently<br>discomforting to<br>interfere with<br>everyday activities | Prevents normal<br>everyday activities<br>or requires medical<br>advice | ER visit or<br>hospitalization |
| Abdominal<br>Pain | None | No interference<br>with activity | Some interference<br>with activity not<br>requiring medical<br>intervention | Prevents daily activity and requires medical intervention | ER visit or hospitalization |
| Anorexia | None | No interference<br>with activity | Some interference<br>with activity not<br>requiring medical<br>intervention | Prevents daily activity and requires medical intervention | ER visit or hospitalization |
| Nausea/<br>Vomiting | None | No interference<br>with activity or 1 to<br>2 episodes/24<br>hours | Some interference with activity or >2 episodes/24 hours | Prevents daily<br>activity, requires<br>outpatient IV<br>hydration | ER visit or<br>hospitalization for<br>hypotensive shock |
| Diarrhea | None | 2 to 3 loose stools<br>or < 400 gms/24<br>hours | 4–5 stools or 400 to 800 gms/24 hours | 6 or more watery<br>stools or ><br>800gms/24 hours or<br>requires outpatient<br>IV hydration | ER visit or<br>hospitalization |
| Malaise/<br>Fatigue | None | No interference with activity | Some interference with activity | Significant; prevents daily activity | ER visit or hospitalization |

<sup>&</sup>lt;sup>a</sup> Everyday activities include attendance at work, school and usual habits of the participants.



**Appendix 2 – Grading of Laboratory Abnormalities (Serum Chemistry)** 

| Serum <sup>a</sup> | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Sodium – Hyponatremia mEq/L | 132 to 134 | 130 to 131 | 125 to 129 | < 125 |
| Sodium – Hypernatremia mEq/L | 144 to 145 | 146 to 147 | 148 to 150 | > 150 |
| Potassium – Hyperkalemia mEq/L | 5.1 to 5.2 | 5.3 to 5.4 | 5.5 to 5.6 | > 5.6 |
| Potassium – Hypokalemia mEq/L | 3.5 to 3.6 | 3.3 to 3.4 | 3.1 to 3.2 | < 3.1 |
| Glucose – Hypoglycemia mg/dL | 65 to 69 | 55 to 64 | 45 to 54 | < 45 |
| Glucose – Hyperglycemia<br>Fasting – mg/dL<br>Random – mg/dL<br>BUN mg/dL | 100 to 110<br>110 to 125<br>23 to 26 | 111 to 125<br>126 to 200<br>27 to 31 | >125<br>>200<br>> 31 | Insulin requirements or<br>hyperosmolar coma<br>Requires dialysis |
| Creatinine – mg/dL | 1.5 to 1.7 | 1.8 to 2.0 | 2.1 to 2.5 | > 2.5 or requires dialysis |
| Calcium – hypocalcemia mg/dL | 8.0 to 8.4 | 7.5 to 7.9 | 7.0 to 7.4 | < 7.0 |
| Calcium – hypercalcemia mg/dL | 10.5 to 11.0 | 11.1 to 11.5 | 11.6 to 12.0 | > 12.0 |
| Magnesium – hypomagnesemia mg/dL | 1.3 to 1.5 | 1.1 to 1.2 | 0.9 to 1.0 | < 0.9 |
| Phosphorous – hypophosphatemia mg/dL | 2.3 to 2.5 | 2.0 to 2.2 | 1.6 to 1.9 | < 1.6 |
| CPK – mg/dL | 1.25 to 1.5 x ULN | 1.6 to 3.0 x ULN | 3.1 to 10 x ULN | > 10 x ULN |
| Albumin – Hypoalbuminemia g/dL | 2.8 to 3.1 | 2.5 to 2.7 | < 2.5 | |
| Total Protein – Hypoproteinemia g/dL | 5.5 to 6.0 | 5.0 to 5.4 | < 5.0 | |
| Alkaline phosphate – increase by factor | 1.1 to 2.0 x ULN | 2.1 to 3.0 x ULN | 3.1 to 10 x ULN | > 10 x ULN |
| Liver Function Tests – ALT, AST increase by factor | 1.1 to 2.5 x ULN | 2.6 to 5.0 x ULN | 5.1 to 10 x ULN | > 10 x ULN |
| Bilirubin – when accompanied by any increase in Liver Function Test increase by factor | 1.1 to 1.25 x ULN | 1.26 to1.5 x ULN | 1.51 to 1.75 x ULN | > 1.75 x ULN |
| Bilirubin – when Liver Function Test is normal; increase by factor | 1.1 to 1.5 x ULN | 1.6 to 2.0 x ULN | 2.0 to 3.0 x ULN | > 3.0 x ULN |
| Cholesterol | 201 – 210 | 211 – 225 | > 226 | |
| Pancreatic enzymes – amylase, lipase | 1.1 to 1.5 x ULN | 1.6 to 2.0 x ULN | 2.1 to 5.0 x ULN | > 5.0 x ULN |

ULN = upper limit of normal

<sup>&</sup>lt;sup>a</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.



Appendix 3 – Grading of Laboratory Abnormalities (Hematology)

| Hematology <sup>a</sup> | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| <u> </u> | | 9.5 to 10.9 | 8.0 to 9.4 | < 8.0 |
| Hemoglobin (Female), gm/dL | 11.0 to 12.0 | 9.5 10 10.9 | 8.0 10 9.4 | < 8.0 |
| Hemoglobin (Female) change from baseline value, gm/dL | Any decrease to<br>1.5 | 1.6 to 2.0 | 2.1 to 5.0 | > 5.0 |
| Hemoglobin (Male), gm/dL | 12.5 to 13.5 | 10.5 to 12.4 | 8.5 to 10.4 | < 8.5 |
| Hemoglobin (Male) change from baseline value, gm/dL | Any decrease to 1.5 | 1.6 to 2.0 | 2.1 to 5.0 | > 5.0 |
| WBC increase, cell/mm <sup>3</sup> | 10,800 to 15,000 | 15,001 to 20,000 | 20,001 to<br>25,000 | > 25,000 |
| WBC decrease, cell/mm <sup>3</sup> | 2,500 to 3,500 | 1,500 to 2,499 | 1,000 to 1,499 | < 1,000 |
| Lymphocytes decrease, cell/mm <sup>3</sup> | 750 to 1,000 | 500 to 749 | 250 to 499 | < 250 |
| Neutrophils decrease, cell/mm <sup>3</sup> | 1,500 to 2,000 | 1,000 to 1,499 | 500 to 999 | < 500 |
| Eosinophils, cell/mm <sup>3</sup> | 650 to 1500 | 1501 to 5000 | > 5000 | Hypereosinophilic |
| Platelets Decreased, cell/mm <sup>3</sup> | 125,000 to<br>140,000 | 100,000 to<br>124,000 | 25,000 to<br>99,000 | < 25,000 |
| PT, increase by factor | 1.0 to 1.10 x ULN | 1.11 to 1.20 x<br>ULN | 1.21 to 1.25 x<br>ULN | > 1.25 ULN |
| PTT, increase by factor | 1.0 to 1.2 x ULN | 1.21 to 1.4 x<br>ULN | 1.41 to 1.5 x<br>ULN | > 1.5 x ULN |
| Fibrinogen increase, mg/dL | 400 to 500 | 501 to 600 | > 600 | |
| | | | | < 100 or |
| Fibrinogen decrease, mg/dL | 150 to 200 | 125 to 149 | 100 to 124 | associated with gross bleeding |
| DIC - disconsinated introversables | | | | or DIC |

DIC = disseminated intravascular coagulation; PT = prothrombin time; PTT = partial thromboplastin time; ULN = upper limit of normal; WBC = white blood cell

<sup>&</sup>lt;sup>a</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.



**Appendix 4 – Grading of Laboratory Abnormalities (Urinalysis)** 

| Urine* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life Threatening (Grade 4) |
|---|---|---|---|---|
| Protein | Trace | 1+ | 2+ | Hospitalization or dialysis |
| Glucose | Trace | 1+ | 2+ | Hospitalization for hyperglycemia |
| Blood (microscopic),<br>red blood cells per<br>high power field | 1 to 10 | 11 to 50 | > 50 and/or<br>gross blood | Hospitalization or packed red blood cells transfusion |

<sup>&</sup>lt;sup>a</sup>The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

Page 27 of 27